CLINICAL TRIAL: NCT03482622
Title: Accurate Assessment of Tumour Clearance During Surgical Treatment of Basal Cell Carcinoma by Fast Raman Spectroscopy
Brief Title: Intraoperative Detection of Residual BCC by Fast Raman
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Nottingham (Other)
Collaborators: Nottingham University Hospitals NHS Trust (Other); Circle Nottingham NHS Treatment Centre (Unknown)
Responsible Party: Sponsor
Other Study IDs: 18003
Record Dates: First submitted 2018-03-14; First posted 2018-03-29 (Actual); Last update posted 2018-03-29 (Actual); Status verified 2018-02

CONDITIONS: Carcinoma, Basal Cell; Intraoperative BCC Detection by Fast Raman Device
Keywords: Raman spectroscopy
MeSH Terms: conditions — Carcinoma, Basal Cell

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients undergoing Mohs surgery: Skin samples excised during Mohs surgery will be measured by the Fast Raman device. The Fast Raman measurements will be compared to gold standard histopathology to determine measurement accuracy.
  Interventions: Diagnostic Test: Fast Raman

INTERVENTIONS:
Diagnostic Test: Fast Raman — Fast Raman uses Raman spectroscopy to measure chemical profiles of tissue and provide a diagnostic map identifying BCC within 30 minutes.

SUMMARY:
The main objective of this research is to develop a new scanning technology called the Fast Raman device, to accurately check the skin removed by the surgeon and detect any residual cancer cells; if found, additional skin can then be removed by surgeons on the same day. The device will be tested first for patients undergoing Mohs micrographic surgery, then be extended to wide-local excisions of basal cell carcinoma (BCC). This study will determine the validity (sensitivity/specificity) and reliability (inter- and intra-user variability) of the Fast Raman device for checking the completeness of tumour removal during Mohs micrographic surgery of BCC.

DETAILED DESCRIPTION:
Raman spectroscopy (RS) is an established analytical technique and has been extensively used in medicine to study individual cells and complex tissues, including skin and skin cancers. This technique is based on inelastic scattering of laser light following its interaction with vibrating molecules of biological samples; therefore, a Raman spectrum represents a "chemical fingerprint" of the sample. Recently, the investigators demonstrated that Raman micro-spectroscopy is able to discriminate between healthy skin and BCC.

With National Institute for Health Research (NIHR) i4i funding (2007-2013), the investigators developed a new technology ("Fast Raman") that can detect BCC regions in skin layers excised during Mohs surgery [13]. A first laboratory prototype based on this technology was able to analyze specimens in 30-60 minutes. In a follow-up i4i project (2014-2016), the investigators have built a fully automated "Fast Raman" device that can be used by non-specialist users and meets the safety requirements to be used in the clinic. The investigators now intend to test this device in real clinical practice and to compare the diagnosis generated by the device with the standard pathology diagnosis.

If the performance of the device achieves the proposed target (~95% sensitivity and specificity, inter-and intra-user reliability higher than typical histopathology, assessment time shorter than frozen section histopathology), it will provide important benefit to BCC patients and health care providers. Faster tissue assessment could speed up Mohs surgery (around 90 mins rather than 3 hours), which is more comfortable for patients. By reducing the costly histopathology procedures needed to process and diagnose skin samples, the Fast Raman device will reduce health care costs, allowing Mohs surgery to become more widely available, and reducing the postcode lottery that currently exists. As the Fast Raman device is designed to be used by non-specialist user, it can be used during any type of BCC surgery, including standard wide local excisions of BCC (>80,000 procedures/year in UK), to provide on the spot an answer on whether the entire tumour has been excised or not.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing Mohs micrographic surgery of BCC.
* Able to give informed consent.
* Any age.

Exclusion Criteria:

* Patients where there is any doubt regarding the diagnosis from pathologist as ascertained by previous diagnostic biopsy.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All consenting patients undergoing Mohs micrographic surgery of BCC.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2018-04-01 (Estimated); Primary Completion 2023-03-31 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
Validity | Immediate
  Accuracy (sensitivity/specificity) of diagnosis made by the Fast Raman device compared to frozen-section histopathology (standard practice) as a the standard of reference.

SECONDARY OUTCOMES:
Reliability | Immediate
  Intra- and inter-user variability in accuracy of Fast Raman results. Identify any conditions (patient groups, tissue types, procedural errors) that cause inaccurate diagnosis.
Measurement Time | Immediate
  Evaluate whether tissue layers can be analysed faster by the Fast Raman device than normal clinical practice.

CONTACTS AND LOCATIONS:
Overall Officials: Ioan Notingher, PhD, Principal Investigator — University of Nottingham

IPD SHARING:
Plan to Share IPD: No
No identifying patient data will be stored as part of this study.

REFERENCES:
- [Derived] Boitor RA, Varma S, Sharma A, Odedra S, Elsheikh S, Eldib K, Patel A, Koloydenko A, Gran S, De Winne K, Koljenovic S, Williams HC, Notingher I. Diagnostic accuracy of autofluorescence-Raman microspectroscopy for surgical margin assessment during Mohs micrographic surgery of basal cell carcinoma. Br J Dermatol. 2024 Aug 14;191(3):428-436. doi: 10.1093/bjd/ljae196. PMID 38736216